CLINICAL TRIAL: NCT06104917
Title: Effect of MaolactinTM Supplement on Gastrointestinal Tract (GIT) Health in Adult Subjects: a Double-blind Randomized Placebo-controlled Study
Brief Title: Effect of Maolactin on Gastrointestinal Tract (GIT) Health
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDC Clinical Pty Ltd (Industry)
Collaborators: Maolac (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAOGIT
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-06

CONDITIONS: Gastrointestinal Dysfunction
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Dose Maolactin (Experimental): Maolactin 500mg per day - 2 capsules containing 250mg active proteins per capsule; equivalent to 500mg active proteins per day
  Interventions: Drug: High Dose Maolactin
- Low Dose Maolactin (Experimental): Maolactin 250mg per day - 1 capsule containing 250mg active proteins per capsule and 1 capsule containing maltodextrin only; equivalent to 250mg active proteins per day
  Interventions: Drug: Low Dose Maolactin
- Maltodextrin (Placebo Comparator): Placebo capsule - 2 capsules containing Maltodextrin per day
  Interventions: Drug: Maltodextrin

INTERVENTIONS:
Drug: High Dose Maolactin — Once daily dose of 2 capsules (2 capsules containing 250mg active proteins per capsule; equivalent to 500mg active proteins per day)
  Arms: High Dose Maolactin
Drug: Low Dose Maolactin — Once daily dose of 2 capsules (1 capsule containing 250mg active proteins per capsule and 1 capsule containing maltodextrin only; equivalent to 250mg active proteins per day)
  Arms: Low Dose Maolactin
Drug: Maltodextrin — Once daily dose of 2 capsules
  Arms: Maltodextrin

SUMMARY:
This is a randomized, double-blind, placebo-controlled, 3 arm parallel group study of 12 weeks duration, with a 4-week run-in period as the control phase and an 8-week intervention period, to investigate the effectiveness of the treatment on upper GI disturbance.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and over
* Generally healthy
* BMI <35kg/m2
* Able to provide informed consent
* Agree to not participate in another clinical trial while enrolled in this trial
* Females using a prescribed form of birth control (e.g. oral contraceptive)
* Experiencing moderate GI disturbances of the upper GI tract - 1 or multiple symptoms (reflux, heartburn, regurgitation, nausea, bloating, abdominal pain) at least once a week for at least 3 months.
* Normal dietary habits (no FODMAP diet, elimination diet, vegan diet, etc) with a minimum 2-month period of self-reported dietary stability.
* Agree to not change current diet and/or exercise frequency or intensity during entire study period
* Agree to not use any dietary supplements for gut health or digestive enzymes during the study period

Exclusion Criteria:

* Unstable(1) or serious illness (e.g. serious mood disorders such as depression or bipolar disorder, neurological disorders such as MS, kidney disease, liver disease, heart conditions, diabetes, thyroid gland dysfunction)
* People with a past or current history of GIT conditions e.g. inflammatory bowel disease, celiac disease or cystic fibrosis as well as gastrointestinal tract surgery
* Current malignancy (excluding BCC) or chemotherapy or radiotherapy treatment for malignancy within the previous 2 years
* Currently taking any proton pump inhibitors [e.g., pantoprazole (Somac), rabeprazole (Pariet), omeprazole (Losec) or any anticoagulation or antiplatelet medications [e.g. Coumadin (Warfarin), Heparin, Dalteparin, Enoxaparin, dabigatran (Pradaxa), rivaroxaban (Xarelto), apixaban (Eliquis), edoxaban (Savaysa), betrixaban (Bevyxxa), clopidogrel (Plavix), prasugrel (Effient), ticagrelor (Brilinta), cilostazol (Pletal) and dipyridamole (Attia, Ofcram, Persantin, Persantin Retard, Trolactin)] including low dose aspirin (acetylsalicylic acid)
* Active smokers, nicotine use or drug (prescription or illegal substances) abuse
* Allergic to any of the ingredients in active or placebo formula
* Pregnant or lactating woman or women trying to conceive
* Any condition which in the opinion of the investigator makes the participant unsuitable for inclusion (including hypercholesterolemia)
* Currently participating in any other clinical trial

Footnote

(1)An unstable illness is any illness that is currently not being treated with a stable dose of medication or is fluctuating in severity. A serious illness is a condition that carries a risk of mortality, negatively impacts quality of life and daily function and/or is burdensome in symptoms and/or treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2025-07-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Change in upper gastrointestinal symptoms | Day -28, Day 0, Day 14, Day 28, Day 56
  Change in upper gastrointestinal symptoms as measured by Gastrointestinal Symptom Rating Scale (GSRS)

SECONDARY OUTCOMES:
Change in upper gastrointestinal symptoms | Day -28, Day 0, Day 14, Day 28, Day 56
  Change in upper gastrointestinal symptoms as measured by Gastroesophageal Reflux Disease Questionnaire (GerdQ)
Change in upper gastrointestinal symptoms | Day -28, Day 0, Day 14, Day 28, Day 56
  Change in upper gastrointestinal symptoms as measured by Bloating Symptoms VAS (BSVAS)
Change in gut microbiome | Day 0, Day 56
  Change in gut microbiome as measured by stool sample analysis
Change in stool frequency and consistency | Day -28, Day 0, Day 14, Day 28, Day 56
  Change in stool frequency and consistency as measured by Bristol Stool Chart
Change in intestinal permeability | Day 0, Day 56
  Change in intestinal permeability as measured by Plasma Zonulin via blood sample
Change in intestinal permeability | Day 0, Day 56
  Change in intestinal permeability as measured by 6 hour urine test
Change in gut inflammation | Day 0, Day 56
  Change in gut inflammation as measured by faecal calprotectin via stool sample
Change in quality of life | Day -28, Day 0, Day 14, Day 28, Day 56
  Change in quality of life as measured by Digestion-associated Quality of Life Questionnaire (DQLQ)
Change in diet | Days -27, -26, -25, Days -3, -2, -1, Days 25, 26, 27, Days 53, 54, 55
  Change in diet as measured by 24-hour Dietary Recall
Change in inflammatory markers | Day 0, Day 56
  Change in inflammation as measured by inflammatory markers (TNFα, interleukin (IL)-1β, IL-6, and IL-8, CRP, Nf-Kb) via blood test
Change in safety | Day 0, Day 56
  Change in safety as measured by E/LFT via including cholesterol and glucose via blood sample
Change in safety | Day -28 to Day 56
  Change in safety as measured by adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- RDC Clinical Pty Ltd, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No